CLINICAL TRIAL: NCT00985257
Title: Performance of the DIDGET Blood Glucose Monitoring System in Children and Young Adults
Brief Title: Performance of a New Glucose Meter System in Children and Young Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ascensia Diabetes Care (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CTD-2009-35
Record Dates: First submitted 2009-09-24; First posted 2009-09-28 (Estimated); Results first posted 2010-11-02 (Estimated); Last update posted 2016-02-29 (Estimated); Status verified 2016-01

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Subjects with diabetes (Other): Subjects with diabetes (or parents/guardians, if applicable)and healthcare professionals (HCPs) use a new blood glucose monitoring system. Subjects were 4 to 24 years of age with type 1 and type 2 diabetes.
  Interventions: Device: DIDGET (Investigational Blood Glucose Monitoring System)

INTERVENTIONS:
Device: DIDGET (Investigational Blood Glucose Monitoring System) — Subjects with diabetes (with parent/guardian assistance, if applicable)and health care professionals (HCPs) each performed duplicate Blood Glucose (BG) tests from the subject's capillary blood on the DIDGET. To test the full range of glucose concentrations, a venipuncture was performed on some subjects to obtain enough blood for modifying (spiking or glycolyzing) to the extreme glucose concentrations. Results were compared to a laboratory glucose method - the Yellow Springs Instrument (YSI) Analyzer.

SUMMARY:
The purpose of this study is to evaluate the performance of a new blood glucose meter in the hands of children, teens, young adults.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 or Type 2 diabetes
* Age 4 to 24 years
* Routinely performs blood glucose testing at home
* If age 18 or older at time informed consent is signed, subject must be able to speak, read, and understand English.
* If younger than age 18, subject's parent/guardian must be able to speak, read, and understand English, and is able to provide appropriate supervision.
* Is willing to complete all study procedures, with or without parent / guardian supervision, if appropriate

Exclusion Criteria:

* Currently pregnant
* Hemophilia or any other bleeding disorder
* Taking prescription anticoagulants (such as Warfarin or heparin) or has clotting problems that may prolong bleeding. Taking Plavix or aspirin daily is not excluded
* Infection with a blood borne pathogen (e.g., HIV, hepatitis)
* Subject or parent/guardian is employee of competitive medical device company
* Cognitive disorder or other condition, which in the opinion of the investigator, would put the person at risk or seriously compromise the integrity of the study

Ages: 4 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 123 (Actual)
Dates: Start 2009-09; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Bailey, MD, Principal Investigator — AMCR Institute; Larry C Deeb, MD PA, Principal Investigator — Larry C. Deeb, MD PA
Locations (2):
- United States (2):
  - AMCR Institute, Escondido, California
  - Larry C. Deeb, MD PA, Tallahassee, Florida

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Subjects With Diabetes
Started | 123
Completed | 123
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Subjects With Diabetes
Number analyzed (Participants) | 123
Age, Customized [Number; unit: participants]
  Age 4-12 years | 41
  Age 13 to 17 years | 30
  Age 18 to 24 years | 52
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69
  Male | 54
Region of Enrollment [Number; unit: participants]
  United States | 123

OUTCOME MEASURES:

1. Primary Outcome: Percent of Blood Glucose (BG) Results Within +/-15mg/dL or +/-20% of Laboratory Glucose Method
Description: Subjects with diabetes and healthcare professionals (HCPs) used a new blood glucose monitoring system (BGMS) with subject blood. BGM results were compared to a lab glucose method - Yellow Springs Instrument (YSI) Analyzer. Duplicate BG results were used to calculate the number of BG results within +/-15mg/dL (for reference BG results <75mg/dL) or +/- 20% (for reference BG values >/=75mg/dL) of the reference method results.
Time Frame: 1-2 hours
Population: To achieve glucose concentrations across the meter test range, 47 blood samples were modified. The total glucose distribution (total 121 natural capillary samples plus 47 modified) ranged from 25.7 to 563.5mg/dL. Two sets of subject results were not analyzed because sufficient sample was not obtained for the YSI reference test.
Measure: Number; unit: percent of blood glucose results
Units Other Than Participants: capillary blood glucose results
Arm/Group | Subjects With Diabetes
Number analyzed (Participants) | 121
Number analyzed (capillary blood glucose results) | 242
percent of blood glucose results
  Subject Tests Natural Capillary n=242=2 x 121 | 97.1
  Combine Natural+Modified n=336=2 x (121+47) | 97.9

ADVERSE EVENTS:
Arm/Group | Subjects With Diabetes
Serious Adverse Events (participants affected / at risk) | 0/123
Other Adverse Events (participants affected / at risk) | 0/123

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less